CLINICAL TRIAL: NCT03020758
Title: The Effect of Bioactives in Dried Plums, Figs, Dates, and Raisins Compared With a High Carbohydrate Snack on Risk Factors for Cardiometabolic Disease
Brief Title: Effect of Dried Fruit on Cardiometabolic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: International Nut and Dried Fruit Council (Unknown); California Dried Plum Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PKE DRIED FRUIT
Record Dates: First submitted 2017-01-03; First posted 2017-01-13 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dried Fruit (Experimental): Daily consumption of ¾ cup blend of dried plums, figs, dates and raisins (DPFDR) for 4 weeks
  Interventions: Dietary Supplement: Dried Fruit
- Control (Experimental): Daily consumption of isocaloric and macronutrient matched snack food for 4 weeks
  Interventions: Other: High Carbohydrate Snack

INTERVENTIONS:
Dietary Supplement: Dried Fruit — Mixture of equal parts 4 dried fruits (figs, raisins, dates, plums) totaling 3/4 cup daily.
  Arms: Dried Fruit
Other: High Carbohydrate Snack — Calorie-matched carbohydrate-rich snack.
  Arms: Control

SUMMARY:
This is a 2-period randomized crossover study with free-living subjects on self-selected diets. The objective of this study is to compare the effects of ¾ cup of a blend of dried plums, figs, dates and raisins (DPFDR) with an isocaloric and macronutrient matched snack food on blood pressure, vascular health and lipids and lipoproteins in 50 participants who are representative of the U.S. population and at risk for cardiovascular disease (overweight/obese, elevated LDL-cholesterol, prehypertension, and/or prediabetes).

The investigators hypothesize that the inclusion of DPFDR in the diet will decrease blood pressure and LDL-cholesterol, and improve artery function (assessed by standard blood pressure measure, 24 hr ambulatory blood pressure, central blood pressure and arterial stiffness) compared to the control group and baseline.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 25-36 kg/m2

And, at least one of the following:

* LDL-C above 116 mg/dL (3.0 mmol/L)
* Systolic blood pressure 120-159 mmHg
* Diastolic blood pressure 80-99 mmHg
* Increased waist circumference: ≥94 cm for men and ≥80 cm for women
* Elevated glucose (≥ 100 mg/dL and < 126 mg/dL)
* Triglycerides: above 150 mg/dL (1.69 mmol/L) and below 350 mg/dL (3.95 mmol/L)
* Low HDL-cholesterol: <40 mg/dL (< 1.03 mmol/L) for men and < 50 mg/dL (<1.29 mmol/L) for women)

Exclusion Criteria:

* Allergies to the test foods
* History of cardiovascular disease, stage II hypertension (BP 160/100 mmHg), kidney disease, diabetes or inflammatory diseases such as gastrointestinal disorders and rheumatoid arthritis
* Use of medication/supplements for elevated lipids, blood pressure, or glucose

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
LDL Cholesterol | 4 weeks
  serum low-density cholesterol concentration

SECONDARY OUTCOMES:
HDL-cholesterol, non-HDL cholesterol, triglycerides | 4 weeks
  serum concentrations of HDL and non-HDL cholesterol and triglycerides
Central blood pressure | 4 weeks
  central systolic and diastolic blood pressure
Pulse wave velocity | 4 weeks
  carotid-femoral pulse wave velocity
Brachial blood pressure | 4 weeks
  brachial systolic and diastolic blood pressure
Plasma glucose | 4 weeks
  fasting plasma glucose
High-sensitivity C-reactive protein | 4 weeks
  serum hs-CRP
Serum insulin | 4 weeks
  fasting serum insulin

OTHER OUTCOMES:
Fecal Microbiome | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Penny Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No